CLINICAL TRIAL: NCT05313971
Title: Impact of Self-awareness in Stress, Burnout, Self-compassion and Compassion in Medical Students - Controlled Clinical Trial
Brief Title: Impact of Self-awareness in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Ines Rosendo, Clinical professor, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 096/2019
Record Dates: First submitted 2022-03-18; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Burnout, Student; Stress, Psychological; Compassion; Self-Perception
MeSH Terms: conditions — Burnout, Psychological; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: After the recruitment period, of the 27 initially enrolled, 24 attended more than 70% of a 28-hour online course, forming the intervention group. The control group was recruited in order to match the age, gender, academic year and teaching faculty variables with the intervention group and people with these characteristics were invited to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 3-week recruitment period of portuguese medical students wanting to attend the 28-hour online course
  Interventions: Other: Self knowledge course
- Control (No Intervention): The control group was recruited in order to match the age, gender, academic year and teaching faculty variables with the intervention group and people with these characteristics were invited to participate.

INTERVENTIONS:
Other: Self knowledge course — The online self-knowledge and communication course, created for the purpose of this clinical trial and taught by professionals with certified training in the area by the Shalom Enneagram Institute (https://iesh.pt/), consisted of providing volunteers with mechanisms for self-knowledge using the enneagram. Three modules were carried out between October and December 2020, spaced in time to allow participants to consolidate knowledge: there was 1 month between the first and second module, and between the second and third, 3 weeks.
  Arms: Intervention

SUMMARY:
Objectives: The goal of this study is to understand whether self-knowledge, using the Enneagram, has a long-term impact as a modifying factor of the quality of life, self-compassion and compassion of medical students.

Methods: An initial sample of 48 medical students answered, before, immediately after and 9 months after an intervention, an online questionnaire with 6 scales. The intervention group took a self-knowledge and communication course based on the Enneagram. The control group was recruited by matching the sociodemographic variables with the intervention group. The data obtained was subject to descriptive and inferential statistical analysis and qualitative content analysis.

DETAILED DESCRIPTION:
Study design Longitudinal study of intervention, controlled, with a reassessment 9 months after the intervention.

Selection of participants The process of recruiting participants involved an online dissemination of the study made by students from the Portuguese Faculties of Medicine of the Universities of Coimbra, Minho, Porto and Lisbon. Interested parties signed up on a Google Form, where the conditions of participation were detailed. The only defined inclusion criterion was to be a medical student enrolled in one of the several Portuguese medical schools.

In order to understand the necessary sample size, the significant results obtained on the Burnout scale of a previous pilot study were used as a basis. The average and the standard deviation obtained before the course and the average achieved after the course of the 3 dimensions of the Burnout scale were inserted into a necessary sample calculation formula, for an alpha of 0.05 and power (1-ß) of 80% (Sample Size Calculator: https://clincalc.com/stats/samplesize.aspx.). We therefore set a target of at least 24 participants needed to form the intervention group.

Data collection Data collection was carried out by filling out a questionnaire on Google Forms lasting about 20 minutes. This collection took place in three stages: both intervention and control groups completed the questionnaire for the first time immediately before the beginning of the first session of the course (phase 1), having repeated it after the conclusion of the third module (phase 2) and again 9 months later (phase 3).

The questionnaire was divided into two distinct parts: the first had the coding of each volunteer for later comparison of data, ensuring their confidentiality, which was followed by the collection of sociodemographic variables: gender, age, academic year and educational institution. The second part was intended to collect the variables of the measured dimensions (perceived quality of life, perceived stress, burnout, self-compassion, compassion and self-reflection and insight), through the application of 6 scales:

1. Visual Analogue Scale for Perceived Quality of Life
2. Perceived Stress Scale
3. Maslach Burnout Scale for Portuguese students
4. Self-Compassion Scale
5. Compassion Scale
6. Self-Reflection and Insight Scale- New Adapted and Validated Self-Awareness Measure for Brazilian Adults In the questionnaires of phases 2 and 3, a last open-response question was added so that the intervention group could share the benefits, in personal terms, in the management of stress and in the relationship and communication with others, which they thought they had acquired with the course.

ELIGIBILITY:
Inclusion Criteria:

* to be a medical student enrolled in one of the several Portuguese medical schools.

Exclusion criteria:

- not participating in 70% of the course (intervention group)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
stress symptoms change | Change from Baseline at 2 months and 11 months
  Perceived Stress Scale (PSS-10: Perceived Stress Scale; Cohen, Kamarck & Mermelstein, 1983 (Cohen et al., 1983); Portuguese version by Trigo et al, 2010) (Trigo et al., 2010). Composed of 10 items, it allows to understand how the unpredictability, uncontrollability or excessiveness of life events are perceived as generators of stress by the individual. Each item is assigned a rating between 0 ("never") and 4 ("very often"). To calculate the final score, it is necessary to reverse the rating of items referring to positive situations (items 4, 5, 7 and 8). Thus, a result between 0 and 40 points is obtained, with values between 0 and 13 being defined as low levels of stress, 14 to 26 medium levels and 27 to 40 high levels. In the Portuguese population, the PSS-10 version has good internal consistency (α=0.87)
burnout risk change | Change from Baseline at 2 months and 11 months
  Maslach Burnout Scale for Portuguese students: Its original version is, to date, the most used burnout rating scale. The version adapted for students (MBI - Student Survey), focusing on feelings and emotions in a school context, comprises 3 subscales, which assess the dimensions Emotional Exhaustion, Disbelief and Professional Effectiveness with 5, 4 and 6 items, respectively. Respondents must rate each of the 15 items between 0 ("never/never") to 6 ("always/everyday"). The final scores are interpreted in the 3 subscales, after the sum of their items, allowing the diagnosis of burnout syndrome when the respondent is simultaneously above the 66th percentile of the Emotional Exhaustion and Disbelief scores and below the 33rd percentile of the Professional Efficacy score, relative to the studied group.
Quality of life change percieved in visual analogue scale | Change from Baseline at 2 months and 11 months
  Visual Analogue Scale for Perceived Quality of Life (EQ-VAS: European Quality of Life - Visual Analogue Scale; EuroQol Group, 1990; Portuguese version by Ferreira, Ferreira & Pereira, 2014) (Ferreira et al., 2013). It is an integral part of the EuroQoL-5Dimension scale (EQ-5D), which comprises two components: a descriptive system, subdivided into 5 dimensions, and a numerical system, achieved through a visual analogue scale - the EQ-VAS thermometer. This offers the possibility for the respondent to quantify their health status on a scale from 0 ("worst imaginable health status") to 100 ("best imaginable health status"), at that moment. In the Portuguese version, the EQ-VAS showed good internal consistency (α=0.862)

SECONDARY OUTCOMES:
compassion change | Change from Baseline at 2 months and 11 months
  Compassion Scale (CS: Compassion Scale; Pommier, 2011 (Pommier, 2011); Portuguese version by Vieira, Castilho & Duarte) (Vieira CS, 2013). Bringing together the six factors of compassion (Kindness vs. Indifference, Common Humanity vs. Disconnectedness, Mindfulness vs. Non-involvement), this scale aims to measure how each individual behaves towards others. Each subject must identify their level of agreement regarding the 24 items of the long version, on a scale from 0 ("almost never") to 5 ("almost always"). Items 1, 2, 3, 5, 7, 10 , 12, 14, 18, 19, 22 and 23, corresponding to subscales with negative connotations (Indifference, Disconnected and Non-Involvement) must be recoded to access the total compassion score. Higher scores translate to a higher level of compassion.
self-compassion change | Change from Baseline at 2 months and 11 months
  Self-Compassion Scale (SELFCS: Self-Compassion Scale; Neff, 2003 (Neff, 2003); Portuguese version of Gouveia & Castilho, 2006) (Castilho & Gouveia, 2011). Considered the most used tool in the assessment of self-compassion, it seeks to measure how the individual behaves in difficult times, through emotional response (Warmness/Understanding vs. Self-criticism), cognitive understanding (Common Humanity vs. Isolation) and attention to one's own suffering. (Mindfulness vs. Overidentification). Each of the 26 items is assigned a rating from 0 ("almost never") to 5 ("almost always"), and it is then possible to calculate the subtotal for each of the six subscales and the total score. For this, all items are summed after recoding items 1, 2, 4, 6, 8, 11, 13, 16, 18, 20, 21, 24 and 25, with higher values reflecting higher levels of self-compassion.
self-reflection and insight change | Change from Baseline at 2 months and 11 months
  Self-Reflection and Insight Scale- New Adapted and Validated Self-Awareness Measure for Brazilian Adults (SRIS: Self-Reflection and Insight Scale; Grant et al., 2002 (Grant et al., 2002); Brazilian version by DaSilveira and DeCastro, 2012) (DaSilveira et al., 2012) ). Self-response instrument with 20 items that seek to assess and measure individual differences in self-awareness, as well as intentional readiness to change behaviour. It contemplates the two-dimensionality of self-awareness through its Insight and Self-reflection subscales, which is subdivided into Need for Self-Reflection and Involvement in Self-Reflection, that is, interest vs. actual execution of the action.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Rosendo, MD PhD, Principal Investigator — Assistant professor FMUC
Locations (1):
- Faculdade de Medicina da Universidade de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
Will not be shared because is not necessary

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05313971/Prot_000.pdf
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05313971/ICF_001.pdf